CLINICAL TRIAL: NCT06673901
Title: Biomechanical Changes in Females with Poly Cystic Ovarian Syndrome
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, rovan mohamed saad elbesh, lecturer, Misr University for Science and Technology
Other Study IDs: NP.T.REC/012/001889
Record Dates: First submitted 2024-09-17; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Poly Cystic Ovarian Syndrome; Polycystic Ovary Syndrome (PCOS)
Keywords: Biomechanical Changes; Spinopelvic alignment; Polycystic Ovarian Syndrome; Hormonal Imbalance; Low-grade Inflammation
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- study group (A): This study enrolled 95 females (52 PCOS, 43 Controls) who agreed to participate in this research. They signed an informed consent after explaining the existence, purpose, and advantages of the study, notifying them of their right to refuse or withdraw at any time. Patients were excluded from the study if they suffered from skeletal deformities (one case), had previous spinal surgeries (one case), had leg length discrepancy (one case) and two cases received hormone replacement therapy
  Interventions: Device: Measurments
- control group (B).: Patients were referred by the gynecologist, based on Rotterdam PCOS Diagnostic Criteria in adults (14), having irregular menstrual cycles (less than 8 menstrual cycles/year or more than 35 days between cycles), painful menses and premenstrual abdominal bloating, and headaches. Forty-three healthy females not suffering from any gynecological condition were referred by a gynecologist and considered the
  Interventions: Device: Measurments

INTERVENTIONS:
Device: Measurments — Each angle was measured three times, and the mean was calculated to represent the data used for statistical analysis. The assessment position for all measurements was relaxed, comfortable standing position and wearing loose clothing, bare feet, and one foot apart between two feet on a level floor in the same room of the same building, at the same time of day. There was a fixed point in the wall, and the woman was instructed to look at it during the assessment; this point adjusts at the level of her eyes. No specific instructions were provided to the females regarding posture so that measurements during a normal standing position. Data was recorded in a data-collecting sheet.
  Other Names: the inclinometer; PALM inclinometer; LH/FSH

SUMMARY:
Polycystic ovarian syndrome (PCOS) is a prevalent endocrine disorder that causes an inversion of the normal luteinizing hormone (LH) to follicle-stimulating hormone (FSH) ratio. Females with PCOS also experience chronic inflammation. This hormonal imbalance and persistent inflammation can reduce muscle strength and mass. Consequently, this may affect the lumbopelvic muscles, potentially leading to postural abnormalities and spinopelvic misalignment.

DETAILED DESCRIPTION:
1.1. Study design This was an observational case-control study. Participants This study enrolled 95 females (52 PCOS, 43 Controls) who agreed to participate in this research. They signed an informed consent after explaining the existence, purpose, and advantages of the study, notifying them of their right to refuse or withdraw at any time. Patients were excluded from the study if they suffered from skeletal deformities (one case), had previous spinal surgeries (one case), had leg length discrepancy (one case) and two cases received hormone replacement therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients were referred by the gynecologist, based on Rotterdam PCOS Diagnostic Criteria in adults (14), having irregular menstrual cycles (less than 8 menstrual cycles/year or more than 35 days between cycles), painful menses and premenstrual abdominal bloating, and headaches.

Exclusion Criteria:

* were excluded from this study if they were obese with BMI > 30 Kg/m2 (obesity induces an increase in anterior pelvic tilt and increased sacral inclination) (15), suffered from musculoskeletal deformities, previous gynecological and spinal surgeries, spinal deformities, leg length discrepancy, orthopedic and neurological disorders, receive hormone replacement therapy (affect functional biomechanical properties by increasing tensile stiffness in the uterosacral ligament and decreasing it in the round ligament)

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: This study enrolled 95 females (52 PCOS, 43 Controls) who agreed to participate in this research. They signed an informed consent after explaining the existence, purpose, and advantages of the study, notifying them of their right to refuse or withdraw at any time. Patients were excluded from the study if they suffered from skeletal deformities (one case), had previous spinal surgeries (one case), had leg length discrepancy (one case) and two cases received hormone replacement therapy
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
I) Pelvic tilt angle | months 6
  While the female was upright, the physiotherapist recorded accurate measurements of the anterior superior iliac spine (ASIS) and posterior superior iliac spine (PSIS). As a result, the therapist adjusted the PALM inclinometer's one end arm on ASIS and the other on PSIS. As detected by the bubble level in the PALM inclinometer, the pelvic sagittal inclination angle was the angle between a horizontal line and a line passing between the ASIS and PSIS. The previous measurement was taken on the right and left sides of the pelvis. This approach has intra-tester solid reliability (ICC = 0.87) and accuracy and validity (17). The mean pelvic tilt angle value ranges from (13° ± 6°)
) Lumbar angle | month 6
  Before the examination, the physiotherapist identifies and applies a skin marker on the spinous processes of the T12 and L5. The inclinometer dial measured the lumbar angle at zero degrees at the wall. Then put the inclinometer kindly but firmly into the inter-spinal spaces at T12 and position at L5, so obtaining the lumbar angle. Neutral values of the lumbar angle are 20º-40º (19). The baseline inclinometer was used with high intra-rater reliability (ICC=0.92) of the bubble inclinometer (20).

SECONDARY OUTCOMES:
LH/FSH | month 6
  Statistical analysis was conducted using SPSS for Windows, version 26 (SPSS, Inc., Chicago, IL). Variances and covariances were homogeneous (p> 0.05), as assessed by Levene's test of homogeneity of variances. Accordingly, parametric statistics were used. Quantitative variables were presented as mean ± standard deviation (X ± SD). An unpaired t-test was used to compare the physical characteristics of both groups. One-way between-subject MANOVA was conducted to determine the differences between both groups in the degree of pelvic inclination, lumbar curve angle, and hormones (LH &FSH). Pearson's correlation coefficient was used to investigate the relationship between pelvic inclination, lumbar curve angle, and hormones (LH &FSH) in females with PCOS. The alpha level was set at 0.05, and the correlation coefficients were interpreted as 0-0.1 = extremely low, 0.10-0.30 = low, 0.30-0.50 = moderate, 0.50-0.70 = high, 0.70-0.90 = extremely high, and 0.90-1.0 = strong

CONTACTS AND LOCATIONS:
Overall Officials: rovan m saad, PHD, Principal Investigator — Misr University for Science and Technology
Locations (1):
- Rovan Elbesh, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided